CLINICAL TRIAL: NCT07204899
Title: Digital Escape Room Game for Hypovolemic Shock Management: A Mixed-Methods Study in Nursing Education
Brief Title: Digital Escape Room Game for Hypovolemic Shock Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, BETUL SAHIN KILINC, Lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17162298600-141
Record Dates: First submitted 2025-06-18; First posted 2025-10-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Nursing Education; Hypovolemic Shock
Keywords: nursing; nursing education; game based learning; digital escape room
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): They were given theoretical training using the traditional method and played a digital escape room game.
  Interventions: Other: Play digital escape room game
- Control group (No Intervention): No intervention was made other than theoretical training using the traditional method.

INTERVENTIONS:
Other: Play digital escape room game — In addition to traditional education, the intervention group will receive a digital escape room game developed with the Genially platform. Both groups' knowledge of Hypovolemic Shock and Nursing Management will be assessed using a fact sheet and satisfaction with the GAMEX scale.
  Arms: Intervention Group

SUMMARY:
Background: Digital escape room games have emerged as innovative pedagogical tools in nursing education, providing immersive and engaging learning experiences. Although their use has expanded to various topics, little is known about their impact in teaching the management of life-threatening emergencies such as hypovolemic shock.

Aim: To evaluate the effects of a digital escape room game on nursing students' knowledge, satisfaction, and perceptions of hypovolemic shock management.

Methods: An explanatory sequential mixed-methods design was employed. In the quantitative phase, a randomized controlled trial was conducted with 55 third-year nursing students assigned to an intervention group (digital escape room) or a control group (traditional lecture). Knowledge levels were assessed at three time points, and the GAMEX scale measured game experiences. In the qualitative phase, focus group interviews were conducted with 12 students from the intervention group to explore experiences in greater depth. Quantitative data were analyzed using repeated-measures ANOVA, and qualitative data were analyzed thematically.

Results: Quantitative findings revealed no statistically significant differences in knowledge scores between the groups over time. However, students in the intervention group reported high levels of enjoyment, motivation, and creative thinking. Qualitative results indicated that the digital escape room reinforced theoretical knowledge, promoted reflection on knowledge gaps, and enhanced critical thinking, problem-solving, and clinical decision-making. Students also emphasized that the game simulated the pressure of real clinical environments, enabling them to practice rapid responses in a safe, engaging context.

Conclusion: Although no significant improvements in knowledge scores were detected, the digital escape room offered substantial educational benefits by strengthening motivation, engagement, and higher-level competencies. It may serve as an innovative complementary strategy to traditional teaching in nursing education.

DETAILED DESCRIPTION:
Study Rationale Traditional lecture-based methods may be limited in preparing nursing students for the complex and time-sensitive decision-making required in managing hypovolemic shock. Digital escape room games provide an immersive, interactive environment where learners collaborate to solve problems under time pressure, simulating aspects of real clinical practice. This innovative format has been applied in various areas of health education, but its impact on teaching emergency management skills such as hypovolemic shock remains underexplored. The present study was designed to evaluate the effectiveness of a digital escape room game in enhancing knowledge, motivation, and higher-order cognitive competencies in nursing students.

Study Design An explanatory sequential mixed-methods design was implemented, combining a randomized controlled trial with a qualitative follow-up phase. The quantitative component compared a digital escape room intervention with a traditional lecture, while the qualitative component explored students' perceptions and experiences in greater depth. This design was selected to capture both measurable outcomes and the underlying mechanisms by which the intervention influenced learning.

Participants Participants were third-year undergraduate nursing students enrolled in a medical-surgical nursing course. A total of 55 students consented to participate and were randomly assigned to either the intervention group (digital escape room) or the control group (lecture). A subsample of 12 students from the intervention arm participated in focus group interviews to provide qualitative insights.

Intervention Model

Experimental Group: Students participated in a digital escape room game specifically developed to teach hypovolemic shock management. The game required students to collaboratively identify clues, apply theoretical knowledge, and make time-pressured decisions to "escape" by stabilizing the patient scenario.

Control Group: Students received a traditional didactic lecture covering the same content on hypovolemic shock management.

Outcome Measures

Primary Outcome: Knowledge of hypovolemic shock, assessed using a structured test administered at three time points (pretest, immediate posttest, and follow-up).

Secondary Outcomes: Learning experiences in the intervention group, assessed using the GAMEX scale, which measures enjoyment, motivation, creative thinking, and other dimensions of game-based learning.

Qualitative Outcomes: Perceptions of the digital escape room's impact on learning, teamwork, and clinical preparedness, explored through thematic analysis of focus group discussions.

Data Collection and Analysis Quantitative data were analyzed using repeated-measures ANOVA to examine changes in knowledge scores over time between groups. GAMEX scores were summarized descriptively. Qualitative data from focus groups were transcribed and thematically analyzed to identify patterns related to perceived learning, challenges, and benefits of the intervention.

Key Findings No statistically significant differences in knowledge scores were observed between the digital escape room and lecture groups. However, students in the intervention group reported high levels of enjoyment, motivation, and creative engagement. Qualitative findings indicated that the digital escape room reinforced theoretical knowledge, revealed knowledge gaps, and fostered critical thinking, problem-solving, and decision-making skills. Students highlighted the game's ability to simulate clinical pressure in a safe, engaging environment.

Conclusion While the digital escape room did not yield significant gains in test-based knowledge, it provided substantial educational value by strengthening learner engagement, motivation, and the development of higher-level competencies. This suggests that digital escape rooms may serve as a valuable complement to traditional teaching strategies in nursing education, particularly in preparing students for the management of emergency clinical conditions such as hypovolemic shock.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 3rd year of the nursing undergraduate program,
* Having signed the voluntary consent form.

Exclusion Criteria:

* Having any health problems that would prevent the continuation of the study, • Requesting to withdraw from the study voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Hypovolemic Shock Information Form to Measure Knowledge Level Regarding Nursing Care in Hypovolemic Shock | On the same day before theoretical training and intervention, 1 day after the intervention and 4 weeks later
  Knowledge of nursing care in hypovolemic shock will be measured using the "Hypovolemic Shock Information Form." A 20-question true-false test was administered to assess students' theoretical knowledge of hypovolemic shock. The minimum possible score on the form is 0, and the maximum is 20. A high score indicates success. To ensure content validity, the form was reviewed by seven field experts and administered as both a pretest and posttest.
GAMEX scale to measure nursing students' satisfaction | on the same day as after the intervention
  Students' experiences with the digital escape room were evaluated using the 27-item, 5-point Likert-type GAMEX scale (Eppman et al., 2018). The instrument comprises six subscales: enjoyment, absorption, creative thinking, involvement, absence of negative effects, and dominance. The Turkish adaptation was validated and found reliable by Arıkan Dönmez et al. (2024). Scale scores range from 27 to 135, with higher scores indicating a more positive gaming experience. Cronbach's alpha was 0.93 for the total scale, and subscale alphas ranged from 0.67 to 0.929.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT07204899/Prot_SAP_001.pdf